CLINICAL TRIAL: NCT07312513
Title: Multicenter, Randomized, Non-inferiority Study to Compare the Performance and Safety of Debrisoft® Duo With Debrisoft® Pad in the Debridement of Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lohmann & Rauscher (Industry)
Collaborators: AXCELLANT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-03
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Ulcers; Arterial Ulcers; Venous Ulcers; Pressure Ulcers; Postoperative Wounds Healing by Secondary Intention; Burns and Scalds; Epidermolysis Bullosa (EB); Traumatic Wounds; Surgical Wounds
Keywords: Debridement; mechanical debridement
MeSH Terms: conditions — Varicose Ulcer; Pressure Ulcer; Burns; Epidermolysis Bullosa; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Debrisoft Duo (Experimental): Patients will be treated with the investigational device which is a two sided pad for the debridement of a wide range of wounds. The soft, wide side of the device is identical to the comparator device. The textured, beige side is unique to the investigational device and makes it easy to loosen strongly adherent, fibrinous wound debris.
  Interventions: Device: two sided debridement pad
- Debrisoft Pad (Active Comparator): Patients will be treated with the comparator device which is a one sided pad for the debridement of a wide range of wounds. The device has the same soft, wide side as the investigational product but does not have the aditional textured, beige side.
  Interventions: Device: one sided debridment pad

INTERVENTIONS:
Device: two sided debridement pad — two sided debridement pad
  Arms: Debrisoft Duo
Device: one sided debridment pad — one sided debridment pad
  Arms: Debrisoft Pad

SUMMARY:
The aim of this post market clinical follow up (PMCF) study is to confirm the performance of Debrisoft® Duo, to collect safety data regarding expected adverse events and to detect potential unexpected adverse events associated with the use of Debrisoft® Duo within the certified indications and under the conditions of routine use.

DETAILED DESCRIPTION:
This clinical investigation will be conducted as multicenter, randomized in parallel groups, non-inferiority controlled trial. After randomization patients will receive wound debrided with the investigational device or the comparator device during one study visit. During the study visit patients will have clinical examination and wound photos will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient is legally capable
* Patient has signed written informed consent
* Presence of one of the following wounds

  * Venous lower leg ulcer
  * Arterial ulcer
  * Diabetic ulcer
  * Pressure ulcer
  * Post-operative wound healing by secondary intention
  * Traumatic wound
  * Surgical wound
  * Burn or scald (grade III: after surgical debridement)
  * Epidermolysis Bullosa
* Wound area >4cm2
* The entire wound area can be displayed on one photo from a distance of 25-30 cm
* Covered with at least 30% debris, necrosis, slough, fibrotic tissue

Exclusion Criteria:

* Known allergy and/or hypersensitivity to Debrisoft® Duo or any of the product components
* Pregnancy or breast feeding
* Patient is illiterate
* Participation in a interventional clinical trial within the last 14 days and during participation in this study
* Any other medical condition, which, by opinion of the investigator, may have impact of the success of the study treatment and/ or interpretation of the study results
* severe pain or hyperesthesia in the wound area
* history of drug or alcohol abuse
* chronic analgesic use (especially opioids) that could influence baseline pain perception
* cognitive impairment, which may affect the ability to accurately self-report pain
* Use of anaesthesia before the debridment procedure
* presence of hard necrotic tissue or other tissue which should not be debrided in general. Other types of hard necrotic tissue requiring debridement, as determined by the investigator, are permitted and may be also pre-moistened before the procedure if deemed necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Relative reduction of fibrinous and necrotic tissue/slough/debris measured by W.H.A.T. | 1 day
  Wound photos will be taken. On these photos, the amount of fibrinous and necrotic tissue/slough/debris in the wound bed before and after debridement will be measured by W.H.A.T. (Wound Healing Analyzing Tool).

SECONDARY OUTCOMES:
Relative reduction of fibrinous and necrotic tissue/slough/debris measured by he investigator | 1 day
  The amount of fibrinous and necrotic tissue/slough/debris in the wound bed before and after debridement will be measured by the investigator.
Rate of device-related adverse events (device safety) | 1 day
  Frequency and character of device deficiencies (DDs), adverse events (AEs), serious adverse events (SAEs), adverse device effects (ADEs), serious adverse device effects (SADEs) and incidents.
Change of wound bed condition, defined by the combination of the following parameters: | 1 day
  * Change in grade of exudate (from very high to none)
  * Change in type of exudate (from haemorrhagic to serous)
  * Change of the wound surrounding skin (presence or abscence of normal, erosive, dry/scaling, dry cracking, oeadematous, red or discoloured skin and cream residues)
  * Change of the wound bed and wound edges (presence or abscence of debris, discoloration, maceration, hyperkeratosis, smooth skin, thickened/rolled edges, undermining, vital tissue, biofilm)
  * Removal of biofilm (estimated by the user)
Wound related pain | 1 day
  Wound related pain will be measured directly before, during and 10 +/-2 minutes using NRS-11 scale
Time needed for debridement | 1 day
  Time needed for the debridement procedure will be assessed using a stopper
Amount of products | 1 day
  Amount of products that were used during one debridement session will be assessed.
Patient satisfaction | 1 day
  Patient satisfaction with the treatment procedure on a scale from 1-5
User satisfaction | 1 day
  User satisfaction assessed via a questionnaire

OTHER OUTCOMES:
Change in wound size | 1 day
  Wound size will be compared before and after the debridement procedure
Results of biopsy or smear | 1 day
  If performed during clinical routine, results of biopsy or smear will be assessed
Removal of biofilm | 1 day
  Change in the presence of biofilm before and after debridement will be investigated using MolecuLightDX. This will only be done at one of the five participating sites.

CONTACTS AND LOCATIONS:
Locations (5):
- Poland (5):
  - MelissaMed Poradnia, Lodz
  - MIKOMED Sp. z.o.o., Lodz
  - NZOZ Neuromed M. i M. Nastaj, Lublin
  - Specjalistyczny Osrodek Leczniczo Badawczy, Ostróda
  - Lecran - Centrum Opieki Nad Ranami-Kunickiego, Wroclaw

IPD SHARING:
Plan to Share IPD: No